CLINICAL TRIAL: NCT00926705
Title: An Intraoperative Infusion of Dexmedetomidine Reduces the Opioid Requirements for Pediatric Patients Undergoing Hypospadias Surgery
Brief Title: Dexmedetomidine Infusion in Hypospadias Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: alghanem2
Record Dates: First submitted 2009-06-22; First posted 2009-06-23 (Estimated); Last update posted 2009-06-23 (Estimated); Status verified 2009-06

CONDITIONS: Pain
Keywords: Dexmedetomidine; Fentanyl; Pain; Pediatrics
MeSH Terms: conditions — Pain | interventions — Dexmedetomidine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fentanyl (Active Comparator): This group received Fentanyl at a dose of 2 ug/kg initially, followed by boluses to keep the patient hemodynamically stable.
  Interventions: Drug: Fentanyl
- Dexmedetomidine and Fentanyl (Experimental): This group received a combination of Dexmedetomidine (1 ug/kg) and Fentanyl (1.79 ug/kg). Total number of patients in this group 24.
  Interventions: Drug: Dexmedetomidine and Fentanyl

INTERVENTIONS:
Drug: Dexmedetomidine and Fentanyl — Dexmedetomidine in a dose of 1 ug/kg initial dose then continuous infusion of 0.7 ug/kg/hr . Combined with Fentanyl at a dose of 2 ug/kg initially plus boluses of fentanyl to keep the patient hemodynamically stable.
  Other Names: Precedex
  Arms: Dexmedetomidine and Fentanyl
Drug: Fentanyl — This group received Fentanyl at a dose of 2 ug/kg initially, followed by boluses to keep the patient hemodynamically stable.
  Arms: Fentanyl

SUMMARY:
The investigators hypothesize that giving Dexmedetomidine in combination with Fentanyl for pediatric patients undergoing hypospadias surgery, will reduce the fentanyl requirement for intraoperative and postoperative analgesia.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-12 years undergoing hypospadias repair

Exclusion Criteria:

* Allergy to Dexmedetomidine
* Preoperative use of sedatives or analgesics
* cardiac diseases
* Children with mental retardation

Ages: 1 Year to 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2008-06; Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Intraoperative and postoperative fentanyl requirement (in microg/kg) | 6/2008-1/2009

CONTACTS AND LOCATIONS:
Overall Officials: Khaled R Al-Zaben, MD, Study Chair — University of Jordan
Locations (1):
- Jordan University Hospital, Amman, Jordan

REFERENCES:
- [Result] Virtanen R, Savola JM, Saano V, Nyman L. Characterization of the selectivity, specificity and potency of medetomidine as an alpha 2-adrenoceptor agonist. Eur J Pharmacol. 1988 May 20;150(1-2):9-14. doi: 10.1016/0014-2999(88)90744-3. PMID 2900154
- [Result] Gurbet A, Basagan-Mogol E, Turker G, Ugun F, Kaya FN, Ozcan B. Intraoperative infusion of dexmedetomidine reduces perioperative analgesic requirements. Can J Anaesth. 2006 Jul;53(7):646-52. doi: 10.1007/BF03021622. PMID 16803911
- [Result] Arain SR, Ruehlow RM, Uhrich TD, Ebert TJ. The efficacy of dexmedetomidine versus morphine for postoperative analgesia after major inpatient surgery. Anesth Analg. 2004 Jan;98(1):153-158. doi: 10.1213/01.ANE.0000093225.39866.75. PMID 14693611
- [Result] Tobias JD, Berkenbosch JW. Sedation during mechanical ventilation in infants and children: dexmedetomidine versus midazolam. South Med J. 2004 May;97(5):451-5. doi: 10.1097/00007611-200405000-00007. PMID 15180019
- [Result] Ibacache ME, Munoz HR, Brandes V, Morales AL. Single-dose dexmedetomidine reduces agitation after sevoflurane anesthesia in children. Anesth Analg. 2004 Jan;98(1):60-63. doi: 10.1213/01.ANE.0000094947.20838.8E. PMID 14693585